CLINICAL TRIAL: NCT05284734
Title: Comparison of Caudal Block and Erector Spinae Block for Postoperative Analgesia in Circumcision and Lower Abdominal Surgery in Pediatric Patients: A Double-blind, Randomized Controlled Trial
Brief Title: Comparison of Caudal Block and Erector Spinae Block for Postoperative Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other)
Responsible Party: Principal Investigator, Volkan Ozen, Associate Professor, Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2021.42
Record Dates: First submitted 2022-03-09; First posted 2022-03-17 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Circumcision; Lower Abdominal Surgery
Keywords: Ultrasound; Pain; Caudal block; Erector spinae block
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Caudal block group (Experimental): A 22 gauge 50 mm echogenic block needle placed through the sacrococcygeal membrane into the sacral canal in the longitudinal position, using the in-plane technique Negative aspiration was then performed 0.125% bupivacaine at a dose of 1 ml/kg was administered
  Interventions: Procedure: Regional anesthesia intervention
- Erector spinae block group (Experimental): The erector spinae muscle and the transverse process were identified, and a 22 G, 80 mm echogenic block needle was advanced towards the transverse process until contact. Following hydrodissection, 1 ml/kg of 0.125% bupivacaine was injected deep into the erector spinae muscle
  Interventions: Procedure: Regional anesthesia intervention

INTERVENTIONS:
Procedure: Regional anesthesia intervention — Ultrasound-guided caudal and erector spinae blocks were administered

SUMMARY:
Caudal block (CB), a regional anesthesia technique, is the most commonly used neuraxial block method for postoperative pain control in sub-umbilical surgeries in children. However, peripheral nerve blocks have been reported to be preferred in recent years in the literature since they provide longer and safer analgesia. One of these blocks, the erector spina plane (ESP) block, has been shown to provide effective postoperative analgesia when administered from the lumbar level for sacral and lower abdominal surgeries and urogenital surgeries in pediatric patients.

DETAILED DESCRIPTION:
Circumcision and any lower abdominal surgery in the pediatric population result in a very painful postoperative period, even when each procedure is evaluated separately. Caudal block (CB), a regional anesthesia technique, is the most commonly used neuraxial block method for postoperative pain control in sub-umbilical surgeries in children. However, peripheral nerve blocks have been reported to be preferred in recent years in the literature since they provide longer and safer analgesia. One of these blocks, the erector spina plane (ESP) block, has been shown to provide effective postoperative analgesia when administered from the lumbar level for sacral and lower abdominal surgeries and urogenital surgeries in pediatric patients. As far as we know, there is no previous study in the literature comparing CB and ESP block in pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* 1-7 years of age
* ASA (American Society of Anesthesiologists) I-II group
* Scheduled for circumcision and unilateral lower abdominal surgery at the same session
* Able to communicate in Turkish
* Willing to participate to the study (parents and children)

Exclusion Criteria:

* Less than 1 or more than 7 years of age
* A neurological deficit, bleeding diathesis, or a history of local anesthetic allergy; an infection or redness in the injection area, congenital lumbar anomaly, liver and/or kidney disorder, a psychiatric disorder, mental retardation, or communication problems detected during examination
* Unwilling to to participate to the study ((parents or children)

Ages: 1 Year to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Level of Postoperative pain | Up to 24 hours
  It was assessed seven times after the operation with Face, Legs, Activity, Cry, Consolability (FLACC) scale. The lowest scale score is 0 points and the highest 10 points.
  Following transfer from the recovery unit to the ward, the 1st, 2nd, 4th, 6th, 12th and 24th hour pain levels were evaluated by the ward nurse.

SECONDARY OUTCOMES:
Time of Postoperative analgesic requirement | Up to 24 hours
  It was assessed seven times after the operation with Face, Legs, Activity, Cry, Consolability (FLACC) scale. The lowest scale score is 0 points and the highest 10 points. Significant pain behavior for the scale has been identified as 4 points or more. Following transfer from the recovery unit to the ward, the 1st, 2nd, 6th, 12th and 24th hour pain levels were evaluated by the ward nurse. Paracetamol was administered IV at a dose of 10 mg/kg if the scale score was 4 or higher.
Rate of Postoperative complications | Up to 24 hours
  Urinary retention, hematoma, ecchymosis, motor block were postoperative complications. They were assessed by an anesthesiologist.

CONTACTS AND LOCATIONS:
Overall Officials: Volkan Özen, Asso.Prof., Principal Investigator — Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Locations (1):
- Prof. Dr. Cemil Tascioglu City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tulgar S, Selvi O, Senturk O, Serifsoy TE, Thomas DT. Ultrasound-guided Erector Spinae Plane Block: Indications, Complications, and Effects on Acute and Chronic Pain Based on a Single-center Experience. Cureus. 2019 Jan 2;11(1):e3815. doi: 10.7759/cureus.3815. PMID 30868029
- [Background] Ozen V, Yigit D. A Comparison of the Postoperative Analgesic Effectiveness of Ultrasound-Guided Dorsal Penile Nerve Block and Ultrasound-Guided Pudendal Nerve Block in Circumcision. Urol Int. 2020;104(11-12):871-877. doi: 10.1159/000509173. Epub 2020 Aug 13. PMID 32791500
- [Background] Ozen V, Yigit D. Caudal epidural block versus ultrasound-guided dorsal penile nerve block for pediatric distal hypospadias surgery: A prospective, observational study. J Pediatr Urol. 2020 Aug;16(4):438.e1-438.e8. doi: 10.1016/j.jpurol.2020.05.009. Epub 2020 May 20. PMID 32507565
- [Derived] Ozen V, Turan EI, Kirdan T, Ayas TA, Erten E, Karacalar S. Erector spinae plane block as an alternative to caudal block in concurrent pediatric urologic and inguinal surgery: A double-blinded randomized controlled trial. Medicine (Baltimore). 2025 Apr 11;104(15):e42109. doi: 10.1097/MD.0000000000042109. PMID 40228275